CLINICAL TRIAL: NCT03016078
Title: A Single Center, Open, Non-controlled Investigation to Evaluate the Performance of a Flexible, Self-adherent Absorbent Silver Dressing Coated With a Soft Silicone Layer After Elective Primary Total Hip or Knee Arthroplasty
Brief Title: Self-adherent Absorbent Silver Dressing in Adults After Hip or Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MxB Po Ag 01
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Arthroplasties, Hip Replacement; Arthroplasties, Knee Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Mepilex Border Post-Op Ag Dressing (Other): A soft silicone foam dressing that absorbs wound exudate maintains a moist wound healing environment and has antimicrobial properties
  Interventions: Device: Mepilex Border Post-Op Ag

INTERVENTIONS:
Device: Mepilex Border Post-Op Ag — To investigate if there was any skin damage under the dressing from operation day to last visit.

SUMMARY:
The overall rationale for this investigation is to evaluate the clinical performance potential for Mepilex Border Post-Op Ag in the ability to minimize the risk of skin related post-operative wound complications such as blistering, maceration and redness at the incision and surrounding skin.

DETAILED DESCRIPTION:
This was a descriptive, open, prospective, non-controlled clinical investigation conducted on 21 enrolled subjects at one site in the United states of America (USA).

The target subjects were male or female, 18 years and older, undergoing elective primary hip or knee arthroplasty with a possibility to participate in a follow-up visit 7 days after surgery. The primary purpose was to investigate if there was any skin damage under the dressing from operation day to last visit. Performance of the dressing as well as comfort, conformability, acceptability and pain at dressing removal was also followed-up until post-op day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Available for a follow-up visit including dressing change 7 days after surgery
3. Plan for elective primary hip or knee arthroplasty
4. Plan for incision size ≤18 cm
5. Provision of informed consent i.e. subject must be able to understand and sign the Patient Information and Consent Form
6. Undergoing elective primary arthroplasty of the hip or knee.

Exclusion Criteria

1. Known allergy/hypersensitivity to any of the components of the dressing
2. Multi-trauma
3. Undergoing arthroplasty due to tumor
4. Previous incision at the same knee or same side of the hip
5. Wound at the surgical site prior to surgery
6. Neurological deficit of operated side (hemiplegia, etc.)
7. Documented skin disease at time of enrollment, as judged by the investigator
8. Previously enrolled in the present investigation
9. Inclusion in other ongoing investigations at present that would preclude the subject from participating in this investigation as judged by the investigator
10. Involvement in the planning and conduct of the clinical investigation (applies to all MHC staff, investigational site staff and third party vendor)
11. Dressing size does not fit the incision area (>18 cm)
12. Complications that would increase wound risks if investigational dressing is applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Myerthall, Dr, Principal Investigator — Center for Orthopedic Research and Education, The CORE Institute
Locations (1):
- The CORE Institute Gilbert, Gilbert, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigation period: Feb 2017 - March 2017. The study was conducted on 21 enrolled subjects at one site in the US. Subjects included were 18 years, and above, undergoing elective primary hip or knee arthroplasty.
Period: Overall Study
Arm/Group | Mepilex Border Post-Op Ag Dressing
Started | 21
Completed | 19
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All variables measured at baseline were summarised for the ITT and PP populations using appropriate summary statistics.
Arm/Group | Mepilex Border Post-Op Ag Dressing
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21
Blistering [Number; unit: Number of blisters] | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Damage to the Incision and Surrounding Skin
Description: The primary outcome is damage to the incision and surrounding skin from operation day to last visit in terms of:
  * Blistering (Yes/No) by visit
  * Redness under dressing (Yes/No) by visit
  * Redness outside dressing (Yes/No) by visit
  * Maceration under dressing (Yes/No) by visit
  * Maceration outside dressing (Yes/No) by visit
Time Frame: Daily visits, up to 7 days
Population: The ITT population included all subjects who underwent at least one post-enrolment treatment. The number of participants analyzed varies due to that no data was captured at some visits, since the dressing was not changed at all visits.
Measure: Count of Participants; unit: Participants
Groups:
- The Study Group: Only one arm. The target subjects were male or female, 18 years and older, undergoing elective primary hip or knee arthroplasty.
Arm/Group | The Study Group
Number analyzed (Participants) | 21
Participants
  Blistering visit 3: number analyzed (Participants) | 1
  Blistering visit 3 | 0
  Blistering visit 5: number analyzed (Participants) | 3
  Blistering visit 5 | 0
  Blistering visit 6: number analyzed (Participants) | 20
  Blistering visit 6 | 0
  Redness Under Dressing visit 3: number analyzed (Participants) | 1
  Redness Under Dressing visit 3 | 0
  Redness Under Dressing visit 5: number analyzed (Participants) | 3
  Redness Under Dressing visit 5 | 0
  Redness Under Dressing visit 6: number analyzed (Participants) | 20
  Redness Under Dressing visit 6 | 5
  Redness Outside Dressing visit 3: number analyzed (Participants) | 1
  Redness Outside Dressing visit 3 | 0
  Redness Outside Dressing visit 5: number analyzed (Participants) | 3
  Redness Outside Dressing visit 5 | 0
  Redness Outside Dressing visit 6: number analyzed (Participants) | 20
  Redness Outside Dressing visit 6 | 2
  Maceration Under Dressing visit 3: number analyzed (Participants) | 1
  Maceration Under Dressing visit 3 | 0
  Maceration Under Dressing visit 5: number analyzed (Participants) | 3
  Maceration Under Dressing visit 5 | 0
  Maceration Under Dressing visit 6: number analyzed (Participants) | 20
  Maceration Under Dressing visit 6 | 0
  Maceration Outside Dressing visit 3: number analyzed (Participants) | 1
  Maceration Outside Dressing visit 3 | 0
  Maceration Outside Dressing visit 5: number analyzed (Participants) | 3
  Maceration Outside Dressing visit 5 | 0
  Maceration Outside Dressing visit 6: number analyzed (Participants) | 20
  Maceration Outside Dressing visit 6 | 0

2. Secondary Outcome: Number of Participants With Leakage of the Dressing
Description: Nurse/ Investigator evaluate: Leakage (No/Yes)
Time Frame: Daily visits, up to 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Study Group
Number analyzed (Participants) | 21
Participants
  Leakage visit 2 | 0
  Leakage visit 3: number analyzed (Participants) | 20
  Leakage visit 3 | 0
  Leakage visit 5: number analyzed (Participants) | 20
  Leakage visit 5 | 0
  Leakage visit 6: number analyzed (Participants) | 20
  Leakage visit 6 | 0

3. Secondary Outcome: Number of Participants With Dressing Sticking to the Staples/Sutures
Description: Nurse/ Investigator evaluate: Dressing sticks to the staples/sutures (No/Yes)
Time Frame: Daily visits, up to 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Study Group
Number analyzed (Participants) | 21
Participants
  Dressing sticks to the staples visit 3: number analyzed (Participants) | 1
  Dressing sticks to the staples visit 3 | 0
  Dressing sticks to the staples visit 5: number analyzed (Participants) | 3
  Dressing sticks to the staples visit 5 | 0
  Dressing sticks to the staples visit 6: number analyzed (Participants) | 20
  Dressing sticks to the staples visit 6 | 0

4. Secondary Outcome: Number of Participants With Bleeding Caused by Dressing Removal
Description: Nurse/ Investigator evaluate: Bleeding caused by dressing removal (No/Yes)
Time Frame: Daily visits, up to 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Study Group
Number analyzed (Participants) | 21
Participants
  Bleeding caused by the dressing removal visit 3: number analyzed (Participants) | 0
  Bleeding caused by the dressing removal visit 3 | 0
  Bleeding caused by the dressing removal visit 5: number analyzed (Participants) | 0
  Bleeding caused by the dressing removal visit 5 | 0
  Bleeding caused by the dressing removal visit 6: number analyzed (Participants) | 2
  Bleeding caused by the dressing removal visit 6 | 0

5. Secondary Outcome: Participants' Dressing Wear Time (Days)
Description: The number of days the dressing can stay on are evaluated
Time Frame: 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | The Study Group
Number analyzed (Participants) | 21
days | 6.35 (1.57)

6. Secondary Outcome: Number of Dressing Changes Per Subject
Description: To evaluate the number of dressing changes per subject
Time Frame: Daily visits, up to 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of dressing changes per subject
Arm/Group | The Study Group
Number analyzed (Participants) | 21
Number of dressing changes per subject | 1.00 (0.00)

7. Secondary Outcome: Evaluation of the Dressing Capacity of Handling Blood
Description: Nurse or Investigator evaluate: Poor, Good, Very Good,Very Good, Excellent on a Likert scale.
Time Frame: Daily visits, up to 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Study Group
Number analyzed (Participants) | 21
Participants
  Poor visit 3: number analyzed (Participants) | 1
  Poor visit 3 | 0
  Poor visit 5: number analyzed (Participants) | 3
  Poor visit 5 | 0
  Poor visit 6: number analyzed (Participants) | 20
  Poor visit 6 | 0
  Good visit 3: number analyzed (Participants) | 1
  Good visit 3 | 0
  Good visit 5: number analyzed (Participants) | 3
  Good visit 5 | 0
  Good visit 6: number analyzed (Participants) | 20
  Good visit 6 | 0
  Very good visit 3: number analyzed (Participants) | 1
  Very good visit 3 | 0
  Very good visit 5: number analyzed (Participants) | 3
  Very good visit 5 | 0
  Very good visit 6: number analyzed (Participants) | 20
  Very good visit 6 | 0
  Excellent visit 3: number analyzed (Participants) | 1
  Excellent visit 3 | 0
  Excellent visit 5: number analyzed (Participants) | 3
  Excellent visit 5 | 3
  Excellent visit 6: number analyzed (Participants) | 20
  Excellent visit 6 | 19
  Not applicable visit 6: number analyzed (Participants) | 20
  Not applicable visit 6 | 1

8. Secondary Outcome: Residuals of the Dressing Material in the Wound or Surrounding Skin at Any Visit (for Patients With at Least One Dressing Change)
Description: Residuals of the dressing material in the wound or surrounding skin at any visit (for patients with at least one dressing change).
  Nurse/ Investigator evaluate with No/Yes
Time Frame: Daily visits, up to 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Study Group
Number analyzed (Participants) | 21
Participants | 3

ADVERSE EVENTS:
Time Frame: Average of one Week
Arm/Group | The Study Group
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Study Group (N=21)
Redness at border of derssing (Skin and subcutaneous tissue disorders) | 1 (1) — Study subject had a distinctive border of redness where the silicone border was present. Subject denied any itching or pain at the incision site, but the PI confirmed it was an AE with a possible relation ADE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03016078/Prot_SAP_000.pdf